CLINICAL TRIAL: NCT05675033
Title: Serplulimab Combined With Anti-VEGF Antibody and Platinum-based Chemotherapy in Treat-naive EGFR/ALK-negative Advanced Lung Adenocarcinoma, a Single Arm Clinical Trail
Brief Title: Serplulimab Combined With Anti-VEGF Antibody in Advanced Lung Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCOG004
Record Dates: First submitted 2022-12-06; First posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-12

CONDITIONS: Lung Adenocarcinoma; Stage IV Non-small Cell Lung Cancer; PD-1 Inhibitor; VEGF
MeSH Terms: conditions — Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Platinum Compounds

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study arm (Other): This is a single arm study.
  Interventions: Drug: Serplulimab and Bevacizumab injection

INTERVENTIONS:
Drug: Serplulimab and Bevacizumab injection — Serplulimab, 4.5mg/kg, intravenous injection, D1,Q21, until the disease progressed or showed intolerable side effects.
  Bevacizumab injection, 7.5mg/kg, intravenous injection, D1, Q21, until the disease progressed or showed intolerable side effects.
  Platinum-based chemotherapy: pemetrexed combined with carboplatin, D1-2, Q21, a total of 4 cycles.
  Other Names: platinum-based chemotherapy

SUMMARY:
In order to further evaluate the efficacy of immunotherapy combined with antivascular therapy in the real world, we used Serpluimab combined with Bevacizumab and platinum-based chemotherapy in previously untreated EGFR/ALK-negative advanced non-squamous NSCLC patients, to evaluate the efficacy and safety of this regimen.

ELIGIBILITY:
Inclusion Criteria:

* Fully understood this study and voluntarily signed the informed consent form (ICF);

  -≥ 18 years and ≤ 75 years old;
* ECOG score 0-1;
* Non-squamous NSCLC;
* stage IV;
* EGFR and ALK negative;
* Treatment-naive;
* According to RECIST1.1 criteria, there are measurable or evaluable lesions.

Exclusion Criteria:

* Tumor histology or cytology confirmed that it was associated with squamous cell carcinoma or small cell lung cancer;
* Patients with severe organ dysfunction were indicated by examination, Exclude subjects with any active, known or suspected autoimmune diseases;
* The estimated survival time is less than 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-10 (Estimated); Primary Completion 2023-01-10 (Estimated); Study Completion 2024-01-10 (Estimated)

PRIMARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  progression-free survival

SECONDARY OUTCOMES:
ORR | up to 12 months
  overall response rate
DCR | up to 12 months
  disease control rate
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | up to 24 months
  Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment